CLINICAL TRIAL: NCT06691776
Title: FASCINATE: FeASibility of Cbct-guIded oNline Adaptive radioThErapy
Brief Title: Feasibility of CBCT-Guided Online Adaptive Radiotherapy (FASCINATE)
Acronym: FASCINATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N23FAS
Record Dates: First submitted 2023-07-13; First posted 2024-11-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Cervical Cancer; Bladder Cancer; Lung Cancer; Head and Neck Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Uterine Cervical Neoplasms; Urinary Bladder Neoplasms; Lung Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized basket trial of the technical feasibility and safety of new software/technologies for CBCT-guided online adaptive radiotherapy. Patients will be enrolled in multiple parallel cohorts, each defined by tumor type(s), and a technical design for the online adaptation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Adapt to rotation for prostate and elective lymph node irradiation (Experimental): The CBCT will be matched (translated and rotated) to the original planning CT with the clinical image registration software. A new software (the rotation simulator) reads both the match of the bony anatomy and the match of the prostate. This software also imports the original planning CT and structures and deforms the original planning CT to match the rotations and translations of pelvis and prostate, as seen in the CBCT. Both these new radiotherapy planning structures and the deformed planning CT are exported to the radiotherapy planning software (Monaco) and used to calculate the adaptive plan. This newly calculated plan will be exported to Mosaiq to treat the patient.
  Interventions: Device: online CBCT-guided adaptive radiation therapy using a new software
- CBCT-guided online adaptation for cervical cancer and elective lymph node irradiation (Experimental): The CBCT will be matched (translated and rotated) to the original planning CT with the clinical image registration software. With in-house software, the target areas and the OARs will be deformed to or segmented on the anatomy of the CBCT. These adjusted radiotherapy structures are then send to the radiotherapy planning software (Monaco). There, the structures are visually inspected and, if needed, manually adjusted. Afterwards, Monaco calculates a new, online adaptive radiotherapy plan. After checking, the plan is exported to Mosaiq to treat the patient.
  Interventions: Device: online CBCT-guided adaptive radiation therapy using a new software
- CBCT-guided online adaptation for bladder cancer. (Experimental): The CBCT will be matched (translated and rotated) to the original planning CT with the clinical image registration software. With in-house software, the target areas and the OARs will be deformed or segmented to the anatomy of the CBCT. These adjusted radiotherapy structures are then send to the radiotherapy planning software (Monaco). There, the structures are visually inspected and, if needed, manually adjusted. Afterwards, Monaco calculates a new, online adaptive radiotherapy plan. After checking, the plan is exported to Mosaiq to treat the patient.
  Interventions: Device: online CBCT-guided adaptive radiation therapy using a new software
- CBCT-guided online adaptation for lung cancer (Experimental): The CBCT will be matched (translated and rotated) to the original planning CT with the clinical image registration software. The rotation simulator reads both the registration of the primary tumor and of the lymph nodes (via the carina). This software also imports the original planning CT and structures and deforms the original planning CT to match the rotations and translations of the primary tumor and lymph nodes, as seen in the CBCT. Both these new radiotherapy planning structures and the deformed planning CT are exported to the radiotherapy planning software (Monaco) and used to calculate the adaptive plan. This newly calculated plan will be exported to Mosaiq to treat the patient.
  Interventions: Device: online CBCT-guided adaptive radiation therapy using a new software
- CBCT-guided online adaptation for head and neck cancer (Experimental): The CBCT will be matched (translated and rotated) to the original planning CT with the clinical image registration software. The rotation simulator reads the image registration of the primary tumor and the match of the lymph node areas. This software also imports the original planning CT and structures and deforms the original planning CT to match the rotations and translations of the primary tumor and lymph node areas, as seen in the CBCT. Both these new radiotherapy planning structures and the deformed planning CT are exported to the radiotherapy planning software (Monaco) and used to calculate the adaptive plan. This newly calculated plan will be exported to Mosaiq to treat the patient.
  Interventions: Device: online CBCT-guided adaptive radiation therapy using a new software

INTERVENTIONS:
Device: online CBCT-guided adaptive radiation therapy using a new software — Patients are treated in the NKI with CBCT-guided online adaptive radiotherapy. While in the clinical workflow one planning CT is used to make the radiotherapy plan, this study treatment creates a new radiotherapy plan on the day of every treatment fraction. Instead of directly irradiating, the radiotherapy plan is adjusted to the anatomy of the day.

SUMMARY:
The accuracy of radiotherapy can be increased by correcting for geometric uncertainties and changes between radiotherapy fractions. These corrections are currently done with online adaptive treatment on a specialized linear accelerator (linac) for a small subset of patients. However, patients currently treated on a standard linac could also benefit from online adaptive radiotherapy. The objective is to determine the feasibility of online CBCT-guided adaptive radiation therapy on a standard Elekta linac.

ELIGIBILITY:
General Inclusion Criteria:

* Patient, age ≥ 18 years, referred for a radiotherapy schedule as described in one of the cohorts.
* WHO performance score 0-3.
* Provision of signed, written and dated IC prior to any study specific procedures.

Specific inclusion criteria for prostate cohort:

* Accepted for radiotherapy of the prostate and pelvic lymph node areas.
* Pathology-proven prostate cancer.
* cT1-4
* cN1 on PSMA-PET/CT or pN1 based on node biopsy, SN-procedure or lymph node dissection.
* cM0 on PSMA-PET/CT (except for patients with M1a disease who are still considered for radiotherapy of the prostate and pelvic lymph node areas).

Specific inclusion criteria for cervical cohort:

* Accepted for radiotherapy of the cervix (with or without chemotherapy) and pelvic lymph node areas (25 fractions, followed by either a brachytherapy or external radiotherapy boost).
* Pathology-proven cervical cancer.
* FIGO IIA2, IB3 and > 6cm, IIB-IVA or N+. Or other stage and unfit for surgery.
* cM0 or cM1 and accepted for locoregional radical (chemo)radiation in 25 fractions.

Specific inclusion criteria for bladder cohort:

* Accepted for radiotherapy of the bladder, either to the entire bladder or with a boost to the tumor area (with or without chemotherapy).
* Pathology-proven bladder carcinoma.
* cT1-4
* cN0 or cN1-2 after induction treatment (with or without lymph node dissection)

Specific inclusion criteria for lung cohort:

* Accepted for radiotherapy for lung cancer with lymph node metastases (with or without chemotherapy).
* Non-small cell lung cancer (either pathology proven or enough clinical suspicion to warrant radiotherapy to primary tumor and pathologic lymph nodes.
* cT1-4 and cN1-3.
* M0 or m1 and accepted for radical radiotherapy in 24 fractions of 1 or more lymph node metastases and a primary tumor and/or pulmonary metastases.

Specific inclusion criteria for head and neck cohort:

* Accepted for radiotherapy for head and neck cancer (with or without chemotherapy).
* Pathology-proven carcinoma of the pharynx, oral cavity or larynx.
* cT1-4
* cN0-3 and indication for elective neck radiation (either 1 or 2 sides).
* cM0

General Exclusion Criteria:

* Patients who are pregnant.

Specific for prostate cohort:

* Patients with a medical condition that severely compromises CBCT image quality (mainly hip prostheses).
* Severe lower urinary tract symptoms that could make the longer treatment time problematic (according to judgement of treating physician).

Specific for cervical cohort:

- Patients with a medical condition that severely compromises CBCT image quality (mainly hip prostheses).

Specific for bladder cohort:

* Patients with a medical condition that severely compromises CBCT image quality (mainly hip prostheses).
* Severe lower urinary tract symptoms that could make the longer treatment time problematic (according to judgement of treating physician).

Specific for lung cohort:

- Severe pulmonary complaints that could make the longer treatment time problematic (according to judgement of treating physician).

Specific for head and neck cohort:

* Severe complaints that could make the longer treatment time problematic (according to judgement of treating physician).
* Pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: successful application of the online adaptive treatment in 90% of 20 patients | From first fraction until the last fraction, an average of 20-35 fractions
  The adaptive treatment is feasible if the technique is successfully ap-plied in 90% of 20 patients.

SECONDARY OUTCOMES:
Safety: Treatment associated ≥ grade 3 acute toxicity according to the NCI Common Terminology Criteria of Adverse Events (CTCAE version 5.0). | From Baseline until 3 months after the last radiotherapy fraction
  Treatment associated ≥ grade 3 acute toxicity according to the NCI Common Terminology Criteria of Adverse Events (CTCAE version 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No